CLINICAL TRIAL: NCT01117675
Title: A New Telemedicine Approach for Chronic HIV/AIDS Patient Home Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Bioengineering and Telemedicine Unit.Universidad Politécnica de Madrid (Unknown)
Responsible Party: Agata Leon/Physician, Hospital Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Hospital Clinic; Universidad Politecnica Madrid
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infection
Keywords: Telemedicine; Home care; Chronic HIV infection; HIV-infected patients
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Other): Arm I: HIV-infected patients controlled through Virtual Hospital
  Interventions: Other: Virtual Hospital
- Arm II (Other): Arm II: HIV-infected patients controlled through Standard Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Virtual Hospital — A new home care model using a telemedicine system (Virtual Hospital) to care chronic HIV-infected patients
  Arms: Arm I
Other: Standard of Care — Standard of Care
  Arms: Arm II

SUMMARY:
Background: Antiretroviral therapy has changed the natural history of the HIV infection in developed countries becoming a chronic disease. This clinical scenario would need a new approach to control patients, simplifying the follow-up visits and the accessibility to the healthcare professionals. A new home care model using a telemedicine system (Virtual Hospital) was developed.

DETAILED DESCRIPTION:
Stable HIV-infected patients with access to a computer and broadband were randomized to: arm I, patients monitored by Virtual Hospital the first year and arm II patients monitored in the hospital the first year (standard of care). After 1 year of follow up, patients were crossed into the other arm. A "Virtual Hospital" was developed to integrate the control of patient in a multidisciplinary telecare team, allowing the patient to be remotely followed-up by the healthcare professionals through Internet. Virtual Hospital had four main services: Virtual Consultations, Telepharmacy, Virtual Library and Virtual Community. A technical and a clinical evaluation of Virtual Hospital were made.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients (CD4 >250 cells/mm3 during at least the 3 months before inclusion to the study)
* Having access to a computer and to a broadband

Exclusion Criteria:

* HIV infected adults with current therapy failure (defined by detectable viral load on treatment or CD4 cell count < 250 cells/ml)
* Tumors
* Opportunistic infections
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of patients cared through Virtual Hospital | Two years
  The main goals were the definition, development, clinical routine installation and evaluation of a telemedicine service that compares standard care with telecare follow-up for attending stable HIV-infected patients in the chronic phase of their disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Agata Leon, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Caceres C, et al. A telemedicine system for chronic HIV/AIDS patient home care through the Internet. Telemedicine and e-Health 2005; 11: 219-220. Caceres C, et al. A Home Integral Telecare System for HIV/AIDS Patients. Stud Health Technol Inform. 2005;114:23-9. Caceres C, et al. An integral care telemedicine system for HIV/AIDS patients. Int J Med Inform. 2006; 75:638-42.
- [Derived] Leon A, Caceres C, Fernandez E, Chausa P, Martin M, Codina C, Rousaud A, Blanch J, Mallolas J, Martinez E, Blanco JL, Laguno M, Larrousse M, Milinkovic A, Zamora L, Canal N, Miro JM, Gatell JM, Gomez EJ, Garcia F. A new multidisciplinary home care telemedicine system to monitor stable chronic human immunodeficiency virus-infected patients: a randomized study. PLoS One. 2011 Jan 21;6(1):e14515. doi: 10.1371/journal.pone.0014515. PMID 21283736